CLINICAL TRIAL: NCT05548075
Title: Psilocybin in Patients With Fibromyalgia: EEG-measured Brain Biomarkers of Action
Acronym: Psilopain
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 275349; EUPAS48284 (Other: EU PAS Register)
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Psilocybin; Lempel-Ziv Complexity; Psychological Flexibility; Chronic Pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Psilocybin; Self-Help Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fibromyalgia Cohort: *As diagnosed by an appropriate medical professional according to the American College of Rheumatology(ACR) diagnostic criteria
  Interventions: Drug: Psilocybin; Behavioral: Therapeutic support

INTERVENTIONS:
Drug: Psilocybin — Up to 25mg of Psilocybin on 2 occasions.
  Other Names: O-phosphoryl-4-hydroxy-N,N-dimethyltryptamine
Behavioral: Therapeutic support — Psychological and physical therapeutic support

SUMMARY:
The purpose of this study is to assess brain activity under Psilocybin in a cohort of people with fibromyalgia.

DETAILED DESCRIPTION:
This mechanistic (Non-CTIMP) study will utilise a within-subjects design to examine a candidate brain biomarker of increased plasticity under Psilocybin. Up to 25mg of Psilocybin will be administered under standardised conditions on two occasions, separated by four weeks with in-dosing EEG recordings.

The primary end-point will take place 8 weeks from the first dosing session after which patients will be remotely monitored monthly for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia lasting for more than 3 months, as diagnosed by an appropriate medical professional using the American College of Rheumatology diagnostic criteria.
* Over 18 years of age
* United Kingdom (UK) resident registered with a primary care medical practice
* Sufficiently competent in English with capacity to provide written informed consent
* Agreement for research team to contact primary and/or secondary care team over the course of the study
* No psychedelic use in the past 6 months

Exclusion Criteria:

* Current or previously diagnosed psychotic disorder or bipolar disorder
* Immediate family member with a diagnosed psychotic disorder
* History of serious suicide attempts or presence of significant suicide/self-harm risk at screening
* Emotionally unstable personality, history of mania, or other psychiatric problem that the screening clinician feels may jeopardise the therapeutic alliance and/or safe exposure to psilocybin
* Currently using medication which could interact with psilocybin including anti-psychotics, mood stabilizers & serotonergic antidepressants including selective serotonin reuptake inhibitors (SSRIs), SNRIs, and tricyclic antidepressants (TCAs)*
* On waiting list for interventional treatment for pain (e.g. surgery or targeted injections)
* Actively enrolled on pain management programme over course of study or awaiting further investigations for pain
* Contraindications to EEG components of the study (e.g., epilepsy, migraine, focal scalp sensitivity)
* MRI contraindications (e.g. claustrophobia, metal implants)
* Physical co-morbidities that are unsuitable for the psychedelic component of the study (e.g., epilepsy, severe cardiovascular disease, insulin-dependent diabetes, hepatic or renal failure e.g., CrCl < 30ml/min etc)
* Blood or needle phobia
* Positive pregnancy test at screening or during the study
* People who are breastfeeding
* Unable to engage with physical demands of dosing session (i.e. attend centre and remain in research facility for an extended period of time)
* Unable to access virtual meetings/phone for remote follow-ups
* Patients consuming more than 35 units of alcohol per week.
* Presence of new or un-investigated 'red flag' symptom indicating need for urgent investigation (e.g. upper motor neuron syndrome, gait ataxia, bladder or bowel dysfunction).
* Limited life expectancy (<18 months) or rapidly deteriorating condition that may inhibit completion of the study (6 month remote follow up).
* Currently prescribed any of the following drugs: Antiepileptics, 5HT3-receptor antagonists, Aspirin, Coumarins, Cyproheptadine, Dabigatran, Dapoxetine, Duloxetine, Lithium, Methylphenidate, Methylthioninium, Metoclopramide, NSAIDs (should be avoided), Naratriptan, Pimozide, Rasagiline, Ritonavir, St John's Wort and Vortioxetine. Tramadol and Fentanyl will be avoided due to their serotonergic action, but all other opioids will not be grounds for exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fibromyalgia lasting for more than 3 months, as diagnosed by an appropriate medical professional using the American College of Rheumatology diagnostic criteria.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Lempel-Ziv complexity (LZc) | 8 weeks
  Lempel-Ziv complexity (LZc) of spontaneous brain activity recorded via EEG.
The Brief Experiential Avoidance Questionnaire (BEAQ) | 8 weeks
  Experiential avoidance as a part component of psychological flexibility

SECONDARY OUTCOMES:
MRI | 8 weeks
  Structural and functional magnetic resonance imaging
Patient reported outcome measures | 6 months
  Secondary outcomes will aim to capture broad aspects of the pain experience
Physiology: Heart rate, body temperature, accelerometry | 8 weeks
  Wearable technology will capture physiological outcomes
Qualitative interviews | 6 months
  Semi-structured and unstructured interviews

CONTACTS AND LOCATIONS:
Overall Officials: David Nutt, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided